CLINICAL TRIAL: NCT07367282
Title: A Phase IV, Prospective, Open-label, Single-arm Clinical Trial to Evaluate the Efficacy of Faricimab and Biomarker Assessment in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Evaluate the Efficacy of Faricimab in Patients With Neovascular Age-related Macular Degeneration
Acronym: nAMD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Junyeop Lee (Other)
Responsible Party: Sponsor-Investigator, Junyeop Lee, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD_ML46106
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Macular Degeneration
Keywords: Neovascular Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — faricimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Faricimab (Experimental): Faricimab injection
  Interventions: Drug: Faricimab Injection [Vabysmo]

INTERVENTIONS:
Drug: Faricimab Injection [Vabysmo] — Faricimab Injection 6mg 0.05 cc

SUMMARY:
If the subject who has nAMD voluntarily agrees to participate in this clinical study by signing the informed consent form, screening assessments will be conducted within 4 weeks prior to the first dose of the investigational drug. During the screening visit, the eligibility of the subject will be assessed and one study eye will be selected. If both eyes are eligible, the eye with the worst best-corrected visual acuity (BCVA) at screening will be chosen. However, if the investigator determines that the other eye requires more urgent treatment for clinical reasons, that eye may be selected as the study eye.

After screening assessments and evaluation based on inclusion/exclusion criteria, eligible subjects will be enrolled. Vabysmo® 6 mg (0.05 mL) will be administered via intravitreal injection every 4 weeks (monthly) for a total of 4 doses during the initial loading period. After the loading dose, patients will undergo disease activity assessment based on imaging and visual acuity (VA) outcomes followed by the IP administration at Week 20. The treatment interval will be determined based on disease activity assessed at Week 20, depending on the results, the subsequent administration may be scheduled at Week 28 or Week 32, at the investigator's discretion. Thereafter, the dosing interval may be further adjusted in 4-week increments, either extended or shortened, according to imaging and visual outcomes.

Throughout the clinical study, patients will need to visit the study site at least 10 times, including the screening visit. The number of intravitreal injections administered will be 4 doses during the initial loading period and up to 5 doses during the treat-and-extend (T&E) period (Weeks 20, 28, 36, 44, 52). Thus, the total number of injections during the study will range from a minimum of 7 to a maximum of 9 injections.

If the non-study eye also has nAMD, treatment with a locally approved therapy may be administered outside the scope of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who voluntarily agree to participate in this clinical study and provide written informed consent
2. Male or female adults aged 50 years or older at the time of consent
3. Individuals who, in the opinion of the investigator, are capable of complying with the requirements of the study protocol

Ocular Conditions

1. Individuals with a BCVA equivalent of ETDRS 24 letters or more, as measured at the time of screening.
2. Confirmed diagnosis, by the investigator, of active nAMD based on sufficiently clear ocular media and adequate pupillary dilation allowing acquisition of good quality retinal images for confirmation.
3. Treatment naïve patients
4. For PCV patients, presence of active polypoidal lesions in the macula as shown by Indocyanine green angiography (ICGA) AND presence of serosanguinous maculopathy
5. For PCV patients, greatest liner dimension (GLD) of the total lesion area <5400 μm as delineated by ICGA.

Exclusion Criteria:

1. Any major illness or major surgical procedure within 1 month before screening.
2. Any condition that, in the opinion of the investigator, constitutes a contraindication to the use of faricimab, may affect interpretation of study results, or places the participant at high risk for treatment-related complications, based on medical history, non-diabetic metabolic abnormalities, physical examination findings, or past/current clinical laboratory results.
3. History of active cancer within 12 months prior to screening, except for adequately treated carcinoma in situ of the cervix, non-melanoma skin cancer, or prostate cancer with a Gleason score ≤6 (Grade Group 1) and stable PSA levels for >12 months.
4. Uncontrolled blood pressure, defined as systolic >180 mmHg and/or diastolic >100 mmHg while at rest at baseline. A repeat reading within the screening window may be taken to confirm eligibility.
5. Immune system abnormalities that may affect inflammatory biomarkers in aqueous humor (AH).
6. History of severe allergic or anaphylactic reaction to biologic agents, or known hypersensitivity to any component of the faricimab injection, study-related procedures (including fluorescein and indocyanine green dyes), dilating drops, or any anesthetic/antimicrobial eye drops used during the study.
7. Systemic treatment for suspected or active systemic infection at screening. Ongoing prophylactic antibiotic use may be acceptable at the investigator's discretion.
8. Use of systemic medications known to have toxic effects on the lens, retina, or optic nerve within 6 months prior to screening or within 5 drug half-lives (whichever is longer), or expected future use of such medications.
9. Receipt of systemic immunomodulatory therapy or immunosuppressive agents within 6 months prior to screening or within 5 drug half-lives (whichever is longer).
10. Participation in another clinical study involving an investigational drug, investigational device, or other medical research within 3 months prior to screening, or concurrent participation in such a study.
11. Pregnant or breastfeeding women.
12. Women of childbearing potential planning to become pregnant during the study or within 3 months after the last dose of study treatment, or unwilling to use highly effective contraception methods* throughout the study period and for 3 months following the last dose.

Ocular Conditions

1. Any ocular condition in the study eye that may interfere with the assessment of visual acuity, safety evaluation, or fundus imaging (e.g., advanced cataract).
2. Any current ocular disease in the study eye that, in the opinion of the investigator, increases the procedural risk of intravitreal injection beyond standard expectations or may interfere with injection, efficacy, or safety evaluations.
3. Presence of fibrosis or atrophy involving ≥50% of the total lesion area and/or the fovea in the study eye, as determined by the investigator.
4. Presence of retinal pigment epithelial (RPE) tear involving the macula in the study eye.
5. High myopia with spherical equivalent refractive error >6 diopters in the study eye. For participants with a history of refractive or cataract surgery, pre-surgical refractive error must not have exceeded -6 diopters.
6. Presence of vitreous hemorrhage in the study eye at screening or baseline visits.
7. History of other macular diseases in the study eye that are unrelated to nAMD but may lead to visual loss or cause intraretinal fluid (IRF) or subretinal fluid (SRF).
8. History or clinical evidence of proliferative diabetic retinopathy, diabetic macular edema, or other retinal vascular diseases in the study eye, other than AMD.
9. Any current ocular condition in the study eye (e.g., cataract) that, in the opinion of the investigator, may require medical or surgical intervention during the study period.
10. History of prior intraocular surgery in the study eye, including but not limited to vitrectomy, glaucoma surgery, corneal transplant, radiation therapy, retinal detachment repair (e.g., scleral buckle or pneumatic retinopexy), trabeculectomy, or other filtration surgeries.
11. History of prior or ongoing treatment for macular neovascularization (MNV) or vitreomacular interface abnormalities in the study eye, including but not limited to intravitreal therapy (faricimab, other anti-VEGF agents, corticosteroids, tissue plasminogen activator, ocriplasmin, C3F8 gas, air), periocular pharmacological interventions, argon laser photocoagulation, verteporfin photodynamic therapy, diode laser, transpupillary thermotherapy, or ocular surgical procedures.
12. Presence of glaucoma in the study eye with uncontrolled intraocular pressure ≥25 mmHg despite pharmacological therapy.
13. Presence of active ocular inflammation or suspected or active ocular or periocular infection in either eye at screening.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
ANG-2 level in aqueous humour (AH) | at Week 20 from baseline
  Measurement of ANG-2 levels in aqueous humor (AH) and the change from baseline to week 20

SECONDARY OUTCOMES:
Endothelial ANG-2 level in aqueous humour (AH) | At weeks 4, 12, 20 and 52 from baseline
  Changes of endothelial ANG-2 level in aqueous humour (AH) at visits compared from baseline at Weeks 4, 12, 20 and 52
BCVA measurement | At weeks 20 and 52 from baseline
  Best Corrected Visual Acuity (BCVA) change from baseline at Weeks 20 and 52
Subfoveal choroidal thickness | At weeks 20 and 52 from baseline
  Change in subfoveal choroidal thickness at Weeks 20 and 52 compared to baseline (limited to PCV patients)
Central subfield thickness (CST) | At weeks 20 and 52 from baseline
  Central subfield thickness (CST) change from baseline at Weeks 20 and 52
Intraretinal microaneurysms and vessel density of the deep capillary plexus | At weeks 20 and 52 from baseline
  Change in the number of intraretinal microaneurysms and vessel density of the deep capillary plexus at Weeks 20 and 52 compared to baseline
Area of peripheral non-perfusion in the retina | At weeks 20 and 52 from baseline
  Change in the area of peripheral non-perfusion in the retina at Weeks 20 and 52 compared to baseline
High improvement in vascular stabilization | from baseline at Weeks 20
  Proportion of patients who achieved high improvement in vascular stabilization at Week 20 (defined as 2 or more score in Macular Neovascularization Stabilisation Scoring System Score range 0-4, higher scores mean a better outcome)
Complete polyp regression | At weeks 20 and 52 from baseline
  Proportion of subjects who experienced complete polyp regression at least once by Weeks 20 and 52 compared to baseline (limited to PCV patients)
Polyp inactivation | At weeks 20 and 52 from baseline
  Proportion of subjects who experienced polyp inactivation at least once by Weeks 20 and 52 compared to baseline (limited to PCV patients)
Resolution of central Intraretinal fluid/Subretinal fluid(IRF/SRF) | At weeks 20 and 52 from baseline
  Proportion of subjects with resolution of central IRF/SRF at Weeks 20 and 52 compared to baseline
Vascular remodeling | At weeks 20 and 52 from baseline
  Proportion of subjects who experiences vascular remodeling with changes in choroidal angiographic features at Weeks 20 and 52 compared to baseline
Number of injections per patient | From baseline to Week 52(EOS)
  Mean number of injections per patient
Treatment interval | From baseline to Week 52(EOS)
  Proportion of subjects who achieved a treatment interval of ≥12 or 16 weeks at least once during the Treat & Extend period
Maximum treatment interval | From baseline to Week 52(EOS)
  Distribution of maximum treatment interval during the Treat & Extend period

OTHER OUTCOMES:
AH biomarkers and imaging biomarkers | From baseline to Week 52(EOS)
  Correlation between AH biomarkers and imaging biomarkers
AH biomarkers and the maximum treatment interval | From baseline to Week 52(EOS)
  Correlation between AH biomarkers and the maximum treatment interval achieved during the T&E period

CONTACTS AND LOCATIONS:
Overall Officials: Junyeop Lee, PhD, Study Director — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No